CLINICAL TRIAL: NCT03221049
Title: the Department of Medical Ultrasonics, Third Affiliated Hospital of Sun Yat-Sen University, 600 Tianhe Road, Guangzhou, China.
Brief Title: Radiomics for Diagnosing Liver Diseases and Evaluating Progression
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Rongqin Zheng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: sysu2017
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis B / Liver Space-occupying Lesions / Patients After Ablation
Keywords: diagnosis performance; hepatocellular carcinoma; liver fibrosis; progression
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular; Liver Cirrhosis; Disease Progression | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- chronic hepatitis B patients: ultrasound and radiomics
  Interventions: Diagnostic Test: radiomics
- patients with liver space occupying lesions: ultrasound and radiomics
  Interventions: Diagnostic Test: radiomics
- patients undergo ablation: ablation, ultrasound and radiomics
  Interventions: Diagnostic Test: radiomics

INTERVENTIONS:
Diagnostic Test: radiomics

SUMMARY:
Liver diseases are worldwide problems. liver fibrosis and hepatocellular carcinoma are mostly concerned by clinicians. Radiomcis can improve diagnosis accuracy and evaluate disease progression. Hence,investors try to combine radiomics and ultrasound images together in order to improve diagnosis performances of liver fibrosis, benign and malignant tumor and progression after liver ablations.

DETAILED DESCRIPTION:
Liver diseases are worldwide problems including diffuse hepatitis disease and liver space occupying lesions. Hepatitis B virus infection is the most important one among difuse hepatitis disease. There are 240 million people infected with HBV globally, and more than one-third of these patients (approximately 93 million) live in China. For them, a precise estimation of the degree of liver fibrosis is important for estimation of prognosis, surveillance, and treatment decisions in patients with HBV infection. Hepatocellular carcinoma is usually detected in liver space occupying lesions and leading to third common death of cancer. Hence, precise diagnosis between benign and malignant tumor is of great significance. Many guidelines recommend ablation as first line treatment to small hepatocellular carcinoma, especially to those less than 1mm.

Liver biopsy has been considered the gold standard for assessing liver diseases. However, it is limited because of sample errors, interobserver variability and many complications, such as pain, bleeding and even death. CT/MR are alternative ways with high cost and complications. Ultrasound was a first optional tool to diagnose liver disease. However, there are still some problems remained to solve:first, the diagnosis accuracy of liver fibrosis remained to be improved. Second,the diagnosis performances for distinguishing benign and malignant tumor were poor. Third, there were not objective way to assess progression after liver ablations.

Radiomcis refers to the extraction and analysis of large amounts of image features from medical images. Previous studies showed that it can improve diagnosis accuracy and evaluating disease progression. Hence,we tried to combined radiomics and ultrasound images together in order to improve diagnosis performances of liver fibrosis, benign and malignant tumor and progression after liver ablations.

ELIGIBILITY:
For chronic hepatitis patients to assess liver biopsy

Inclusion Criteria:

* HBsAg positive or HBV-DNA detected
* agreed to undergo liver biopsy
* agreed to participated in our study

Exclusion Criteria:

* combined with other liver disease(eg. HAV/HCV/HDV,alcoholic liver disease)
* combined with HIV
* combined with malignant liver space occupying lesions
* liver transplantation
* pregnant
* the sample size of liver biopsy could not demand: length lower than 15mm, portal areas less than 6.

For patients classified between benign and malignant tumor

Inclusion Criteria:

* patients diagnosed with liver space occupying lesions
* with histology results of liver space occupying lesions.
* agreed to participate in our study and signed informed consent.

Exclusion Criteria:

* ultrasound images cant meet the demand for analysis
* without histology results

For patients to estimate progression after ablation

Inclusion Criteria:

* patients diagnosed with hepatocellular carcinoma;
* patients treated with ablation;
* patients performed the contrast-enhanced ultrasonography before ablation;
* patients who treated with transcatheter arterial chemoembolization (TACE) performed the contrast-enhanced ultrasonography performed before TACE;

Exclusion Criteria:

* patients with lack of US digital imaging data
* loss to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: chronic hepatitis B patients /patients with liver space occupying lesions / patients after ablation
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
liver fibrosis | 1 year
  the degree of liver fibrosis
benign or malignance | 5 years
  the malignance of liver space occupying lesions
The incidence of recurrence | 5 years
  the incidence of liver cancer recurrence after ablation

CONTACTS AND LOCATIONS:
Overall Officials: rongqin zheng, doctor, Principal Investigator — The department of Ultrasound, the third affiliated hospital of Sun Yat-sen University
Locations (1):
- The department of Ultrasound, the third affiliated hospital of Sun Yat-son University, Guangzhou, Guangdong, China